CLINICAL TRIAL: NCT01929811
Title: Neoadjuvant Treatment of TEC Versus TEC Plus Metformin in Breast Cancer：A Prospective, Randomized Trial
Brief Title: NeoMET Study in Neoadjuvant Treatment of Breast Cancer
Acronym: NeoMET
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow enrollment.
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Kunwei Shen, Professor, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RJBC1301
Record Dates: First submitted 2013-08-11; First posted 2013-08-28 (Estimated); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: pCR Rate; BCT Rate; Safety
MeSH Terms: interventions — Metformin; Docetaxel; Epirubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin arm (Experimental): Docetaxel: 75mg/m2, d1, q3w*6 Epirubicin: 75mg/m2, d1, q3w*6 Cyclophosphamide: 500mg/m2, d1, q3w*6 Metformin: 500mg tid, orally (500mg daily in first cycle)
  Interventions: Drug: Metformin; Drug: Docetaxel; Drug: Epirubicin; Drug: cyclophosphomide
- TEC (Other): Docetaxel: 75mg/m2, d1, q3w*6 Epirubicin: 75mg/m2, d1, q3w*6 Cyclophosphamide: 500mg/m2, d1, q3w*6
  Interventions: Drug: Docetaxel; Drug: Epirubicin; Drug: cyclophosphomide

INTERVENTIONS:
Drug: Metformin — Metformin: 500mg tid, orally (500mg daily in first cycle) on day 1 to day 21 of each 21 day cycle
  Other Names: Metformin HCL; Metformin hydroehloride
  Arms: Metformin arm
Drug: Docetaxel — 75 mg/m2, IV (in the vein) on day 1 of each 21 day cycle; 6 cycles.
Drug: Epirubicin — 75 mg/m2, IV (in the vein) on day 1 of each 21 day cycle; 6 cycles.
Drug: cyclophosphomide — 500 mg/m2, IV (in the vein) on day 1 of each 21 day cycle; 6 cycles.

SUMMARY:
To evaluate docetaxel, epirubicin and cyclophosphomide (TEC) with TEC plus metformin in neoadjuvant treatment of breast cancer patients. The aim is to evaluate whether metformin can increase the pCR rate combination with TEC regimen in neoadjuvant setting.

DETAILED DESCRIPTION:
Neoadjuvant therapy is the standard treatment for locally advanced breast cancer and has adopted in early breast cancer treatment. A meta-analysis showed no difference between neoadjuvant therapy and adjuvant therapy in terms of survival and overall disease progression. Therefore, neoadjuvant treatment can be offered as a standard treatment and as an alternative to adjuvant treatment to all patients who are expected to be candidates for adjuvant systemic chemotherapy. Patients achieved pCR after treatment have superior outcome.

The taxanes were introduced into clinical practice in the early 1990s, and recent meta-analysis showed that compared with anthracycline-containing chemotherapy, taxanes-containing regimens significantly reduced the annual breast cancer recurrences and deaths. Right now, TAC regimen has widely accepted as adjuvant or neoadjuvant chemotherapy regimens in breast cancer treatment.

Metformin, an inexpensive oral agent commonly used to treat type 2 diabetes, has been garnering increasing attention as a potential anti-cancer agent. In neoadjuvant treatment of breast cancer, a retrospective clinical study from MDACC reported a significantly increased pCR rates to standard neoadjuvant chemotherapy in diabetic breast cancer patients who were receiving metformin (24% pCR) compared to diabetics not receiving metformin (8% pCR), with intermediate rates in non-diabetics who did not receive metformin (16% pCR), indicating metformin may increase pCR rate with neoadjuvant chemotherapy.

Base on these data, we initiate a prospective study to evaluate docetaxel, epirubicin and cyclophosphomide (TEC) with TEC plus metformin in neoadjuvant treatment of breast cancer patients. Our aim is to evaluate whether metformin can increase the pCR rate combination with TEC regimen in neoadjuvant setting.

ELIGIBILITY:
Inclusion Criteria:

* women aged ≥18 years and < 70 years with life expectancy > 12 months
* Measurable disease in breast or axillary lymph node, histologically confirmed invasive breast cancer by core needle biopsy, T≥2cm or stage IIb or stage III according AJCC classification, fine-needle aspiration is encouraged to every patient with metastasis suspicious nodes;
* Biopsy specimens are available for ER, PgR, Her2 and proliferation biomarker detection;
* Adequate bone marrow function: Neutrophil ≥ 1.5*109/L; Hb ≥ 100g/L; PLT ≥ 80*109/L;
* Adequate liver and renal function:
* Serum AST ≤ 90U/L
* Bilirubin ≤ upper limit of normal (UNL) range
* Serum creatinine ≤110 umol/L，calculated creatinine clearance should be ≥ 60 mL/min;
* BUN ≤ 7.1mmol/L;
* Has ECOG Performance Score 0-1;
* BMI ≥ 25kg/m2 or hyperglycemia or hyperlipemia or hypertension;
* Willing to take biopsy before neoadjuvant chemotherapy and patients must be accessible for treatment and follow-up;
* Women with potential child-bearing must have a negative pregnancy test (urine or serum) within 7 days of drug administration and agree to use an acceptable method of birth control to avoid pregnancy for the duration of the study;
* Written informed consent according to the local ethics committee requirements.

Exclusion Criteria:

* Prior systemic or loco-regional treatment of breast cancer, including chemotherapy;
* Metastatic breast cancer;
* With a history of malignant tumor except uterine cervix cancer in situ or skin basal cell carcinoma;
* Patients with medical conditions that indicate intolerant to neoadjuvant therapy and related treatment, including uncontrolled pulmonary disease, severe infection, active peptic ulcer, coagulation disorder, connective tissue disease or myelo-suppressive disease;
* Has active hepatitis B or hepatitis C with abnormal liver function tests (LFTs) or is known to be HIV positive;
* Contraindication for using dexamethasone, chemotherapy agents or metformin;
* History of congestive heart failure, uncontrolled or symptomatic angina pectoris, arrhythmia or myocardial infarction; poorly controlled hypertension (systolic BP >180mmHg or diastolic BP >100mmHg);
* Has peripheral neuropathy ≥ grade 1;
* Patient is pregnant or breast feeding (not willing to stop breast feeding);
* Not willing to take core needle biopsy or patients with psychiatric disorder or other diseases leading to incompliance to the therapy
* Known severe hypersensitivity to any drugs in this study;
* Treatment with any investigational drugs within 30 days before the beginning of study treatment.
* History of lactic or other metabolic acidosis
* Consumption of > 3 alcoholic beverages per day (on average)

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
pathologic complete response rate | 5 months
  To compare pathologic complete response (pCR) rate to neoadjuvant chemotherapy between Docetaxel, Epirubicin and Cyclophosphamide (TEC) arm and TEC plus Metformin arm in breast cancer.
  Definition of pCR is no invasive tumor in primary breast and axillary lymph node.

SECONDARY OUTCOMES:
Clinical response rate | up to 4.5 months
  To compare the clinical response rate between Docetaxel, Epirubicin and Cyclophosphamide (TEC) arm and TEC plus Metformin arm in breast cancer neoadjuvant treatment.
safety profile | up to 4.5 months
  To compare the tolerability and side effects of neoadjuvant chemotherapy between Docetaxel, Epirubicin and Cyclophosphamide (TEC) arm and TEC plus Metformin arm in breast cancer treatment.
breast conservation therapy (BCT) rate | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Kunwei Shen, Dr., Principal Investigator — Ruijin Hospital
Locations (2):
- China (2):
  - Linyi People's Hospital, Linyi, Shandong
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality

REFERENCES:
- [Derived] Huang J, Tong Y, Hong J, Huang O, Wu J, He J, Chen W, Li Y, Chen X, Shen K. Neoadjuvant docetaxel, epirubicin, and cyclophosphamide with or without metformin in breast cancer patients with metabolic abnormality: results from the randomized Phase II NeoMET trial. Breast Cancer Res Treat. 2023 Feb;197(3):525-533. doi: 10.1007/s10549-022-06821-y. Epub 2022 Dec 16. PMID 36525180